CLINICAL TRIAL: NCT05944588
Title: Predictive Value of Chest Ultrasound Observation on Extubation Failure
Acronym: ECHOEXTUB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0031
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Ultrasound; Weaning Failure; Ultrasound; Lung Edema; Extubation Failure
Keywords: Extubation; Weaning Failure; Lung Ultrasound; Chest Ultrasound; B Lines
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extubation Success: Patients who don't need a new intubation in the 7 days following the extubation
  Interventions: Other: Pulmonary Ultrasound
- Extubation Failure: Patients who need a new intubation in the 7 days following the extubation
  Interventions: Other: Pulmonary Ultrasound

INTERVENTIONS:
Other: Pulmonary Ultrasound — 2 pulmonary ultrasound exams, one before respiratory weaning test, and one other at the end of the respiratory weaning test, before extubation

SUMMARY:
The use of mechanical ventilation in intensive care concerns the majority of patients, most often to compensate for respiratory failure, but for other organic failures requiring therapeutic artificial coma. During the sedation phase, many elements of management can modify the patient's clinical parameters.

Indeed, mechanical ventilation with a positive expiratory pressure mainly modifies the venous return by decreasing it, and therefore many modifications of the hemodynamic parameters result from it. In addition, other elements of management, such as iterative fillings, vasopressor and inotropic amines, as well as sedative drugs not only modify the hemodynamics, but also the ventilatory mechanics.

Extubate a patient in intensive care is always complex, because the assessment must be multifactorial and this is not without risk for the patient. Many complications can arise if it ends in failure. They can be linked to mechanical causes (laryngeal oedema, tracheal stenosis, pneumothorax...) but also to non-mechanical causes, such as inappropriate sedation, overload, neuromuscular deficit. Extubation is primarily based on the patient's level of consciousness, as well as the successful progress of the patient during a ventilatory weaning trial, carried out after a return to spontaneous ventilation with inspiratory support. This ventilatory weaning test precedes extubation and is performed for any patient intubated for more than 48 hours.

Since the 1950s, ultrasounds have become more and more important in the field of medical diagnosis and therapeutic decision support, even more recently in the world of intensive care. The contribution of echocardiography in a patient in the process of extubation has already been evaluated and has proven to be a valuable aid. For nearly 20 years, the use of pulmonary ultrasound has emerged and allows rapid diagnosis at the patient's bedside of mechanical anomalies such as gaseous or liquid effusion, an anomaly in the compliance of the pulmonary parenchyma, possibly in link with diaphragmatic dysfunction or even signs in favor of a picture of pulmonary overload, thanks to ultrasound artefacts such as B lines or even alveolar derecruitment by atelectasis.

The role of pulmonary ultrasound in helping to decide on extubation remains poorly established, we propose an observational study evaluating the predictive value of chest ultrasound in pre-extubation with the aim of determining if ultrasound signs are able to predict a potential failure of this extubation. Indeed, the risks of extubation failure being much higher than those of ventilatory weaning failure, it seems necessary to focus our research on this component.

This study must include patients in spontaneous mechanical invasive ventilation with pressure support, presenting the criteria for a ventilatory weaning test in view of a potential extubation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with organ failure requiring intubation for more than 48 hours
* In spontaneous ventilation with pressure support
* Presenting the common criteria of the unit to start a ventilatory weaning test
* Richmond Agitation Sedation Scale 0

Exclusion Criteria:

* Sedated patient with a score of 0 at the Richmond Agitation Sedation Scale
* Pregnant woman
* Patient under guardianship or curators or deprived of public rights
* Patient with a contraindication to performing an external ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the intensive care unit of the University hospital of Caen, presenting the Eligibility criteria without any exclusion criteria, intubated since more than 48h, presenting the common criteria of the unit to start a ventilatory weaning test
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-05-22 (Estimated); Study Completion 2024-05-22 (Estimated)

PRIMARY OUTCOMES:
Determine if pulmonary ultrasound observations are predictive factors linked with extubation failure | 7 days
  See if there's more pathological ultrasound signs in the extubation failure group

SECONDARY OUTCOMES:
Determine at wich range of pathological ultrasound observations there's a positive correlation with extubation failure | 7 days
  See if there 's a specific range number of pathological observations, where we can start to see a link with the extubation failure

CONTACTS AND LOCATIONS:
Overall Officials: Damien DD DUCHEYRON, PHD, Principal Investigator — University Hospital Center of Caen
Locations (1):
- University Hospital Center, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: No